CLINICAL TRIAL: NCT05570760
Title: Clinical Study to Evaluate Adaptos®Ortho Wedge Bone Graft Substitute in High Tibial Osteotomy: A Randomized, Controlled, Partially Blinded, Multi-Center Trial.
Brief Title: Clinical Study to Evaluate Adaptos®Ortho Wedge Bone Graft Substitute in High Tibial Osteotomy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biomendex Oy (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AdaptosOrtho-001
Record Dates: First submitted 2022-08-02; First posted 2022-10-07 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Knee Deformity
Keywords: synthetic bone graft; Adaptos; high tibial osteotomy; orthopaedics
MeSH Terms: interventions — Bone Transplantation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

ARMS (3):
- Adaptos®Ortho Wedge (Experimental): Bone augmentation after Open Wedge High Tibial Osteotomy (OWHTO), with Adaptos®Ortho Wedge (Biomendex Oy, synthetic bone graft material) in combination with a load bearing TomoFix® Medial High Tibia Plate (DePuy Synthes).
  Interventions: Device: Adaptos®Ortho Wedge (bone grafting surgery)
- No bone graft (Sham Comparator): OWHTO with unfilled bony defect of the osteotomy gap with a load bearing TomoFix® Medial High Tibia Plate (DePuy Synthes).
  Interventions: Procedure: OWHTO without bone grafting
- chronOS® Wedge (Active Comparator): Bone augmentation, after OWHTO, with chronOS® Wedge (DePuy Synthes, synthetic beta-TCP bone graft) in combination with a load bearing TomoFix® Medial High Tibia Plate (DePuy Synthes).
  Interventions: Device: chronOS® Wedge (bone grafting surgery)

INTERVENTIONS:
Device: Adaptos®Ortho Wedge (bone grafting surgery) — After screening and enrollment, subjects will undergo medial knee open wedge high tibial osteotomy (OWHTO) with load bearing locking plate fixation. A synthetic bone graft will be used as a bone void filler in the osteotomy defect. Follow-up visits will be at 6 weeks, 3 months, 6 months, and 12 months.
  Arms: Adaptos®Ortho Wedge
Procedure: OWHTO without bone grafting — After screening and enrollment, subjects will undergo medial knee open wedge high tibial osteotomy (OWHTO) with load bearing locking plate fixation, without bone grafting. Follow-up visits will be at 6 weeks, 3 months, 6 months, and 12 months.
  Arms: No bone graft
Device: chronOS® Wedge (bone grafting surgery) — After screening and enrollment, subjects will undergo medial knee open wedge high tibial osteotomy (OWHTO) with load bearing locking plate fixation. A synthetic bone graft will be used as a bone void filler in the osteotomy defect. Follow-up visits will be at 6 weeks, 3 months, 6 months, and 12 months.
  Arms: chronOS® Wedge

SUMMARY:
The aim of this study is to obtain performance and safety data of the new investigational device, dual-part Adaptos®Ortho Wedge, for its intended use in orthopaedic surgery. The study intervention is medial open wedge high tibial osteotomy (OWHTO) with loadbearing plate fixation, where a bone graft substitute material Adaptos®Ortho Wedge is evaluated when used as a bone void filler. Investigational device is expected to support bone formation in osteotomy gap and to resorb in the body.

The comparator arms are treated with medial OWHTO with plate fixation, either without a bone graft (the bone defect is left empty, non-augmented osteotomy) or by using a comparator product (chronOS® Wedge, semi-circular) as a bone void filler.

DETAILED DESCRIPTION:
The study aims to evaluate the clinical performance and safety of Adaptos®Ortho Wedge (Biomendex Oy) bone graft material, when used for filling the medial osteotomy gap of the knee during OWHTO surgery.

This is partially randomized, subject and outcome assessor-blinded, controlled, multi-center study. The total study duration for each patient is planned to be 12 months. In total 6 visits per patient are scheduled in this study.

The study has three arms, and patients of all study arms are treated with medial OWHTO surgery to treat unicompartmental medial misalignment of the knee. Participants in the experimental arm (Arm 1) receive the investigational device, the osteotomy gap is filled with Adaptos®Ortho Wedge bone graft substitute. Participants in the control arm (Arm 2) receive the OWHTO treatment, where the osteotomy gap is left empty (no bone graft). Participants in the comparator device arm (Arm 3) receive the OWHTO treatment, where the osteotomy gap is filled with chronOS® Wedge bone graft substitute. In all three groups the metallic fixation plate (TomoFix®) is used for load bearing and for stabilizing the defect. The study device chronOS® Wedge (DePuy Synthes) and TomoFix® (DePuy Synthes) are CE-marked. The products are used within the indication.

The subject will be followed for twelve months following OWHTO.The radiological bone regeneration in the bony defect will be assessed at 6-weeks and 3-, 6-, and 12-months post-surgery.

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged between 25 and 65 years at the time of enrolment.
* Subjects that sign and date a written, informed consent form (ICF) prior to the initiations of any trial procedures, after the nature of the trial has been explained according to regulatory requirements.
* Subjects who can comply with trial procedures and are available for the duration of the trial.
* Accepts all treatment arms.
* Subjects with varus malalignment of the knee, scheduled to have medial open-wedge high tibial osteotomy (OWHTO) but are otherwise in good health at the time of entry into the trial as determined by medical history, physical/clinical examination, and clinical judgement of the investigator.
* Full knee range of motion (ROM) (at least 5-120 degrees).
* Preoperatively planned osteotomy 5-13 degrees of the proximal tibia done based on the weight-bearing x-ray of the full leg in AP view using Miniaci Method.
* Body Mass Index (BMI) ≤30

Exclusion Criteria:

* Previous knee area osteotomy or lower limb arthroplasty of the investigational knee.
* Presence of the following unfavourable conditions: osteoporosis, infectious/inflammatory joint disease, infections, or inflammation in the operation area, clinically relevant, not medically managed, severe acute or chronic medical illness, immune-compromised, metabolic/systemic bone disorder, untreated malignant myeloma, Burkitt's lymphoma, lateral osteoarthritis (Kellgren-Lawrence grade >1)
* Smoking or use of other nicotine products
* Inability to follow the procedures of the study, e.g. due to language problems, dementia, psychiatric disorder or behaviour etc. of the participant
* Recent history of substance abuse (ie, recreational drugs, alcohol) that would preclude reliable assessment.
* Women who are pregnant or breast feeding or planning to become pregnant during the study.
* Any use of calcitonin, bisphosphonates or recombinant PTH 1-34, 1-84 or other PTH fragments/analogues 6 months prior to surgery or during the study (12 months po).
* Enrolment of the investigator, his/her family members, employees, and other dependent persons.
* Involved in study of another investigational product that may affect outcome.

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 87 (Estimated)
Dates: Start 2024-04-08 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Radiographic bone regeneration of the osteotomy defect, comparison between three treatment arms. | Change from baseline to 12 months.
  Radiographic bone regeneration assessments of the native x-ray of the standing anteroposterior (AP) radiographs of the knee, evaluated in the mediolaterally divided five zones of the osteotomized gap area (Brosset 2011), with rating of six bone remodeling phases (phases 0-5, with the score of 5 for the best outcome).The primary endpoint is the sum of the remodeling phase scores (0-5) in each of the five zones of the osteotomized gap area (range 0-25). Assessment longitudinally at 6-weeks and repeatedly at 3-, 6-, and 12-months post-surgery. Primary evaluation is done 12 months after surgery.

OTHER OUTCOMES:
Bone union of the tibial posterior cortex | Change from baseline to 12 months.
  Bone union of the tibial posterior cortex is assessed on lateral radiographs. Assessed at 6 weeks, 3-, 6-, and 12- months post-operation.
Questionnaire: KOOS (Knee Injury and Osteoarthritis Outcome Score) | Change of KOOS score from baseline to 12 months.
  Patient-reported outcome measure (PROM) relating to knee pain and function. KOOS is a 42-item questionnaire. KOOS consists of 5 subscales; Pain, other Symptoms, Function/activities in daily living (ADL), Function in sport and recreation (Sport/Rec) and knee related Quality of life (QOL). Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4. A normalized score (100 indicating no symptoms and 0 indicating extreme symptoms) is calculated for each subscale. Assessed at preoperative visit, and 6 weeks, 3-, 6-, and 12- months post-operation.
Questionnaire: FJS (Forgotten Joint Score) | Change from baseline to 12 months.
  Patient-reported outcome measure (PROM) focusing on patients' awareness of a specific joint in everyday life. FJS is a 12-item questionnaire. When calculating the total score for the FJS, all responses are summed (never, 1 point; almost never, 2 points; seldom, 3 points; sometimes, 4 points; mostly, 5 points) and the raw score is linearly transformed to obtain a total score range of 0 to 100. Finally, the score is subtracted from 100 to change the direction of the final score in such a way that high scores indicate a high degree of "forgetting" the joint-i.e. a low degree of awareness. Assessed at preoperative visit, and 6 weeks, 3-, 6-, and 12- months post-operation.
NRS Knee Pain Intensity score | Change from baseline to 12 months.
  Patient reported outcomes relating to pain. Pain intensity is rated on a numeric rating scale where zero indicated no pain at all, and 10 represented the worst possible pain. Assessed at preoperative visit, and 6 weeks, 3-, 6-, and 12- months post-operation.
Questionnaire: overall satisfaction to the procedure | Change from baseline to 12 months.
  Procedure satisfaction questionnaire. The study subjects complete 5-point Likert scale satisfaction questionnaire. The response category for subjects is 1 (Very dissatisfied), 2 (Dissatisfied), 3 (Neither satisfied nor dissatisfied), 4 (Satisfied), and 5 (Very satisfied). Assessed at 6 weeks, and 3-, 6-, and 12- months post-operation.
Bone union in the defect area | The change from baseline to 12- months post-operation
  Bone union assessed on AP radiographs (+/-) at 6 weeks, and 3-, 6-, and 12-months post-surgery.
Knee CT scan | 6 months post-operation.
  Clinical assessment of bone regeneration, as based on computed tomography (CT) images of the knee.
Full loadbearing | Up to 3 months post-operation.
  The date (or follow-up week, +/- 1 week) when a patient is capable of full loadbearing, to abandon crutches conclusively. Outcome measure will be assessed up to 3 months visit.
Mechanical axis Hip knee ankle angle | The change from baseline to 12- months post-operation.
  The HKA angle in degrees is measured.
Mechanical axis weight-bearing line ratio | The change from baseline to 12- months post-operation.
  The WBL ratio in percentage is measured.
Work disability days | Up to 3 months post-operation.
  The date when a patient returned to work after surgery is recorded (number of work disability days post-surgery). Outcome measure will be assessed up to 3 months visit.

CONTACTS AND LOCATIONS:
Overall Officials: Mikko Manninen, MD, PhD, Study Director — Orton Oy
Locations (6):
- Finland (3):
  - Kanta-Häme Central Hospital, Hämeenlinna
  - Meilahti Bridge Hospital, Helsinki University Hospital, Helsinki
  - Pihlajalinna Kelloportti, Tampere
- Hungary (3):
  - Petz Aladár University Teaching Hospital, Győr
  - University of Szeged Szent-Györgyi Albert Clinical Center, Szeged
  - Szent György University Teaching Hospital, Székesfehérvár

IPD SHARING:
Plan to Share IPD: No